CLINICAL TRIAL: NCT02432950
Title: PANCREATIC NUTRITIONAL PROGRAM (PNP): A Novel Weight Reduction Program in Overweight/Obese Breast Cancer Survivors
Brief Title: Pancreatic Nutritional Program for Weight Loss in Overweight/Obese Patients With Stage I-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14253; NCI-2015-00654 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14253 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Obesity; Breast Neoplasms | interventions — Diet Therapy; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (PNP) (Experimental): Patients participate in the PNP intervention, which begins with a baseline meeting with a diet and lifestyle instructor to discuss baseline testing results, begin an educational plan, determine an individualized eating plan, and print out food choices. Patients also undergo automated glucometry every 15 minutes, review their individual food choices and blood glucose levels 90 minutes after eating, keep a daily nutrition and lifestyle journal log, fill out a daily meal discovery card log, and attend weekly meetings with a diet and lifestyle instructor for 12 weeks.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Participate in the PNP
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Educational Intervention — Participate in the PNP
  Other Names: Education for Intervention; Intervention, Educational
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot clinical trial studies a pancreatic nutritional program for helping patients with stage I-III breast cancer who are overweight or obese lose weight. When patients have a high level of sugar in their blood, due to eating sugary foods and/or a sedentary lifestyle, the pancreas needs to work harder to digest the sugar. This can cause weight gain, obesity, and other illnesses. Breast cancer patients who are overweight and obese are more likely to have their breast cancer return. The pancreatic nutritional program is a diet and lifestyle intervention that helps protect the pancreas by keeping blood sugar levels low, and may help patients achieve sustained weight loss, improved health, better quality of life, and possibly a better outcome to their treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the change in body weight at 6 months post-intervention relative to baseline.

SECONDARY OBJECTIVES:

I. To examine changes in: body composition; body chemistry; physical fitness; inflammatory markers; deoxyribonucleic acid (DNA) repair capacity; and quality of life per the Functional Assessment of Cancer Therapy - Breast (FACT-B)+4, version 4 questionnaire at 6 months post-intervention relative to baseline.

II. To describe adverse events possibly related to wearing the glucometer sensor or following the pancreatic nutritional program (PNP) diet.

III. To document compliance with the various components of the PNP (wearing the glucometer sensor; recording body weight; completing journal entries; completing meal cards; attending weekly counseling sessions with diet instructor).

OUTLINE:

Patients participate in the PNP intervention, which begins with a baseline meeting with a diet and lifestyle instructor to discuss baseline testing results, begin an educational plan, determine an individualized eating plan, and print out food choices. Patients also undergo automated glucometry every 15 minutes, review their individual food choices and blood glucose levels 90 minutes after eating, keep a daily nutrition and lifestyle journal log, fill out a daily meal discovery card log, and attend weekly meetings with a diet and lifestyle instructor for 12 weeks.

After completion of study, patients are followed up within 1 week and then at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early-stage breast cancer (stage I-III)
* Patients who have or have not undergone chemotherapy are both eligible; if the patient has undergone chemotherapy she must have completed adjuvant chemotherapy for >= 3 months and =< 5 years prior to study enrollment
* Postmenopausal women defined by either: natural menopause with at least one year since last menses, or chemotherapy-induced menopause with at least one year since last menses and follicle-stimulating hormone (FSH) and estradiol levels within the postmenopausal range
* Body mass index (BMI) of 25-33 kg/m^2
* Patients must be willing to adhere to the PNP intervention and the entire 6-month study
* All patients must have the ability and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who are diabetic
* Patients whose BMI falls outside the eligible range (< 25 kg/m^2 or > 33 kg/m^2)
* Patients with stage IV breast cancer
* Patients with Rheumatoid Arthritis and other inflammatory diseases that would impact correlative studies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 6 months
  Tested using the paired t-test, alpha = 0.05.

SECONDARY OUTCOMES:
Change in body chemistry (lipid panel; comprehensive metabolic panel; complete blood count; fasting blood glucose; insulin resistance) | Baseline to up to 6 months
  Tested using the paired t-test, alpha = 0.05. P values will not be adjusted for multiple hypothesis testing.
Change in body composition (BMI) | Baseline to up to 6 months
  Tested using the paired t-test, alpha = 0.05. P values will not be adjusted for multiple hypothesis testing.
Change in physical fitness (measured using a handgrip dynamometer) | Baseline to 6 months
  Tested using the paired t-test, alpha = 0.05. P values will not be adjusted for multiple hypothesis testing.
Change in quality of life score (FACT-B+4) | Baseline to 6 months
Change in serum inflammatory markers (C-reactive protein; cytokines) | Baseline to 6 months
  Tested using the paired t-test, alpha = 0.05. P values will not be adjusted for multiple hypothesis testing.
Compliance metrics (days glucometer sensor not utilized; days body weight not recorded; days journal entries not made; days meal cards not created; weekly counseling sessions missed) | 12 weeks
DNA repair capacity (comet assay's mean olive tail moment; number of gamma-H2A histone family, member X foci) | Baseline to 6 months
  Tested using the paired t-test, alpha = 0.05. P values will not be adjusted for multiple hypothesis testing.
Incidence of adverse events reported as possibly or definitely related to wearing the glucometer sensor following the PNP diet | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States